CLINICAL TRIAL: NCT01134354
Title: The Role of Patient Expectations in Traumatic Orthopedic Outcomes TEFTOM: The Trauma Expectation Factor - Trauma Outcomes Measure TEFTOM EURASIA
Brief Title: The Role of Patient Expectations in Traumatic Orthopedic Outcomes-TEFTOM EURASIA
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: TEFTOM EURASIA
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Tibia Fracture (Isolated); Ankle Fracture (Isolated)
Keywords: Validation study; Outcome Measures; Patient Outcomes Assessment; Patient expectations; Physician patient relationship
MeSH Terms: conditions — Tibial Fractures; Ankle Fractures

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TEFTOM: Patient outcome measure

SUMMARY:
Design:

Prediction trial, up to 10 sites in Asia and Europe

Goal:

To better understand the "success" or "failure" after orthopedic trauma surgery by developing a model that can be applied clinically as a user-friendly "baseline" questionnaire - capable of predicting "success" or "failure" based on a patient's pre-surgical expectations of their final outcome and to validate a novel outcomes measure (TOM).

Primary aim:

To assess the psychometric properties of predictive validity, internal consistency and reproducibility of the trauma expectation factor (TEF) in the Eurasian population.

Secondary aim:

To assess the psychometric properties of criterion validity, internal consistency,reproducibility, and sensitivity to change of the TOM in the Eurasian population.

Key questions related to patient and surgeon expectations:

* How different, or similar, are patient and surgeon expectations?
* Do expectations change over time?
* Do patient expectations predict outcomes in validated measures use today?

ELIGIBILITY:
Inclusion Criteria:

* Isolated ankle or distal tibia fracture
* Scheduled for and undergoing one of the following surgeries for their fracture:

  * Open fracture and internal fixation (ORIF)
  * external fixation (EF)
  * EF followed by ORIF
* 18 years of age or older
* Understand and read country national language at elementary level
* Able to understand the purpose of the clinical trial,
* Able and willing to conduct all follow-up visits
* Signed informed consent

Exclusion Criteria:

* Subject has previously undergone internal fixation surgery for this ankle/distal tibia fracture.
* Subject has disease entity, or condition that precludes likelihood of bony union (e.g., metastatic cancer, metabolic bone disease).
* Subject has severe dementia or other severe mental health problem that may preclude him/her from completing study questionnaires.
* Subject is participating in other competing clinical research that may interfere with participation in this research.
* Subject is unlikely to attend study related follow-up visits.
* Subject has poly-trauma (more than one organ system compromised)
* Subject has additional fracture(s) other than ankle fracture
* Subject is a prisoner
* Fracture occurred more than 28 days before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient 18 years of age or older with an isolated ankle or distal tibia fracture, scheduled for and undergoing one of the following surgeries for their fracture (Open fracture and internal fixation (ORIF, external fixation (EF) or EF followed by ORIF)
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2010-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Teftom Questionnaire | one year

CONTACTS AND LOCATIONS:
Overall Officials: Reto Babst, MD, Principal Investigator — Luzerner Kantonsspital
Locations (7):
- China (2):
  - Queen Mary Hospital, Hong Kong
  - Shanghai Sixth People's Hospital, Shanghai
- Universitätsklinikum Köln, Cologne, Germany
- HOSMAT Hospital, Bangalore, India
- Hospital Universitari de Girona Doctor Josep Trueta, Girona, Spain
- Switzerland (2):
  - Kantonsspital Luzern, Lucerne
  - Stadtspital Triemli, Zurich